CLINICAL TRIAL: NCT03308539
Title: Predictive Value of Epicardial Fat Thickness for Disease Severity in Coronary Artery Disease Patients
Brief Title: Prediction of Coronary Artery Disease Severity by Epicardial Adipose Tissue Thickness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Osama Fekry (Other)
Responsible Party: Sponsor-Investigator, Osama Fekry, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: epicardial adipose tissue
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myocardial infarction patients: transthoracic echocardiography and cardiac magnetic resonance
  Interventions: Radiation: echocardiography and cardiac magnetic resonance

INTERVENTIONS:
Radiation: echocardiography and cardiac magnetic resonance — transthoracic echocardiography and magnetic resonance imaging of the heart

SUMMARY:
is to test the hypotheses that epicardial adipose tissue can be a marker of severity of coronary artery disease in myocardial infarction patients

DETAILED DESCRIPTION:
epicardial adipose tissue is defined as the adipose tissue between the visceral pericardium and the outer margin of the myocardium which can be considered an endocrine organ that secretes pro-inflammatory and anti-inflammatory cytokines and chemokines including adiponectin.as investigators know, inflammatory response is an important factor in the coronary atherogenesis. Therefore,epicardial adipose tissue is likely to be connected with the severity of coronary artery disease.Recent studies showed that the thickness of the epicardial adipose tissue in patients with coronary artery disease was greater than that with normal coronary arteries.

epicardial adipose tissue will be assessed using transthoracic echocardiography and cardiac magnetic resonance which allows for an accurate volumetric quantification of epicardial fat.

ELIGIBILITY:
Inclusion Criteria

1. Normal thoracic shape
2. Sinus rhythm
3. without severe respiratory diseases

Exclusion Criteria:

1. contraindication for cardiac magnetic resonance.
2. Patients who previously underwent coronary artery bypass grafting or percutaneous coronary angiography prior to admission
3. history of chronic kidney disease with glomerular filtration rate <30 mL/min
4. pericardial and/or pleural effusion.

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: acute myocardial infarction patiens not previously underwent percutaneous coronary angiography or coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
measurement of epicardial adipose tissue as marker of severity of coronary artery disease in myocardial infarction patients. | one year
  epicardial adipose tissue measurement using transthoracic echocardiography and cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- Jacqueline George, Asyut, Single, Egypt

REFERENCES:
- [Result] Desferrioxamine and transfusional iron overload. Lancet. 1978 Mar 4;1(8062):479-80. No abstract available. PMID 76025